CLINICAL TRIAL: NCT07239791
Title: Role of the Noradrenergic System in the Regulation of Learning Dynamics: Evaluation of the Effect of a Low-dose Selective Noradrenaline Reuptake Inhibitor (NOISYXETINE)
Acronym: NOISYXETINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D24-P017
Record Dates: First submitted 2025-09-29; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Role of the Noradrenergic System in the Regulation of Learning Dynamics; No Disease or Condition is Being Studied
Keywords: noradrenaline; learning dynamics; atomoxetine; healthy subject
MeSH Terms: interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Single centre, double-blinded, randomized, placebo-controlled, cross-over study involving 160 evaluable healthy adults. Subjects will be separated in 2 cohorts: A for participants having the stable task and B for those having the changing one. They will then be randomized in a 1:1 ratio to one of the 2 treatment sequences:
  * Atomoxetine 40 mg - Placebo (Subgroups A1 or B1);
  * Placebo - Atomoxetine 40 mg (Subgroups A2 or B2).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Atomoxetine 40 mg - Placebo (Other): The participants will receive one cap of atomoxetine 40 mg at V1 and placebo at V2
  Interventions: Drug: Atomoxetine; Drug: Placebo
- Sequence 2: Placebo - Atomoxetine 40 mg (Other): The participants will receive one cap of placebo at V1 and atomoxetine 40 mg at V2
  Interventions: Drug: Atomoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — One single capsule of atomoxetine 40 mg given at one visit according to the sequence randomly allocated.
  Placebo of atomoxetine will be administered at the other visit for the participant (according to the sequence randomly allocated)
Drug: Placebo — One single capsule of placebo given at one visit according to the sequence randomly allocated.

SUMMARY:
Administration of low-dose selective noradrenaline reuptake inhibitor (sNRI) (e.g. atomoxetine) to healthy subjects is a validated model of increasing cortical noradrenaline levels which, combined with computational modelling of behaviour, allows fine-grained analysis of the impact on learning processes of noradrenaline's fluctuations in the human cortex.

The study goal is to characterize the modifications of certain cognitive processes and associated brain circuits under low-dose sNRI using validated computational learning models. The study will be interested in how subjects will modify their learning under the effect of the drug across two separate investigations; one utilizing in a stable evidence accumulation task and one utilising a changing evidence accumulation task. This approach will help to better understand the link between noradrenaline and accumulation of evidence in healthy subjects, and indirectly in some neuropsychiatric pathologies.

The study is a single centre, double-blinded, randomized, placebo-controlled, cross-over study involving evaluable healthy adults separated in 2 cohorts: A for participants having the stable task and B for those having the changing one. Participants will then be randomized in a 1:1 ratio to one of the following treatment sequences:

* Atomoxetine 40 mg - Placebo (Subgroups A1 or B1);
* Placebo - Atomoxetine 40 mg (Subgroups A2 or B2).

DETAILED DESCRIPTION:
Hundred and sixty healthy volunteers will be enrolled (80 / task) in 24 months. The maximum duration of participation for each subject is 51 days.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed, assessed by the Edinburgh scale;
* Written signed informed consent;
* Subject covered by a social security regimen.

Exclusion Criteria:

* Pregnant, parturient or breastfeeding woman;
* First-degree family history of axis I disorder (DSM-IV-TR), excepted unipolar mood and anxiety disorders with OCD;
* Personal history of axis I disorder (DSM-IV-TR) in the 6 months preceding the study entry;
* Dependence on a psychoactive substance in the 12 months preceding the study entry, excluding nicotine, any behavioural disorder incompatible with a 2-hour electroencephalographic recording;
* Neuro/psychotropic treatment ongoing or stopped less than 1 month ago;
* Personal history of neurological pathology (e.g.: congenital malformation, benign or malignant tumour, degenerative disease of the central nervous system (CNS), epilepsy, inflammatory or infectious disease of the CNS, etc.);
* Personal history of chronic disease of infectious, neoplastic, vascular, dysimmune or inflammatory, metabolic or endocrine, degenerative or genetic aetiology. In particular, angle-closure glaucoma, pheochromocytoma, known high blood pressure or measured blood pressure greater than 140/90 mm Hg at baseline, congenital heart disease, known ischemic heart disease, known heart failure, supraventricular or ventricular heart rhythm disorder, nephropathy, known liver disease and any pathology likely to be aggravated by an increase in blood pressure;
* Any medical treatment in the month preceding the study entry, apart from effective contraceptive treatment;
* Subject deprived of liberty by a judicial or administrative decision;
* Person subject to a legal protection measure or unable to express consent;
* Known intolerance to atomoxetine;
* Need to wear glasses and/or lenses to obtain normal vision;
* Subject in an exclusion period or enrolled in an interventional study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Apparent Learning rate | From Visit 1 (Day 0) to Visit 2 (Day 7)
  Paired difference in the apparent learning rates (in both environmental contexts: stable task and changing task), between the sNRI (atomoxetine) and control (placebo) conditions.
  Apparent learning rate will be calculate with the following formula: αt=(vt- vt-(1) )/(xt- vt-1) according to Foucault and Meyniel (Foucault C, Meyniel F (2024) Two Determinants of Dynamic Adaptive Learning for Magnitudes and Probabilities. Open Mind : Discov Cogn Sci 8:615-638) The learning rate measures the amount of update of the learned value (from vt-(1 to vt) induced by the observation xt in proportion to its deviation from the previously learned value.

SECONDARY OUTCOMES:
Number of adverse events | From Visit 1 (Day 0) to Visit 2 (Day 7)
  Side effects (treatment related adverse events) in all groups between study drug administration at Visit 1 (Day 0) and Visit 2 (Day 7) including vital signs worsening and ECG findings
Change from Visit 1 (Day 0) in the computational modelling of behaviour at Visit 2 (Day 7) | From Visit 1 (Day 0) to Visit 2 (Day 7)
  Computational modelling of behaviour at Visit 1 and 2: paired difference in latent behavioral parameters of the computational models that characterize the learning process (in a stable accumulation task and in a dynamic accumulation task), between the sNRI (atomoxetine) and control (placebo) conditions.
Change from Visit 1 (Day 0) in the score of the State Trait Anxiety Inventory (STAI) questionnaire at Visit 2 | From Visit 1 (Day 0) to Visit 2 (Day 7)
  The scores of the State Trait Anxiety Inventory (STAI) questionnaire (Spielberger et al., 1983) will be compared between Hour 0 and Hour 3 at Visit 1 and 2 to control for the effect of the substance on the subjects' levels of depression and anxiety.
  The STAI comprises 2 questionnaires of 20 items with the following ranges:
  * STAI-YA (state anxiety): 0-80 with 0 equivalent to no anxiety and 80 the worst possible anxiety
  * STAI-YB (Trait anxiety): 0-80 with 0 equivalent to no anxiety and 80 the worst possible anxiety
Change from Visit 1 (Day 0) in the score of the Beck Depression Inventory (BDI) questionnaire at Visit 2 | From Visit 1 (Day 0) to Visit 2 (Day 7)
  The scores of the Beck Depression Inventory (BDI) questionnaire (Beck et al., 1961) will be compared between Hour 0 and Hour 3 at Visit 1 and Visit 2 to control for the effect of the substance on the subjects' levels of depression.
  The BDI comprises 21 items with the following ranges: 0-63 with 0 equivalent to no depression and 63 the worst possible depression.
Change from Visit 1 (Day 0) in the score of visual analogue scale (VAS) on anxiety at Visit 2 | From Visit 1 (Day 0) to Visit 2 (Day 7)
  The scores of the VAS-anxiety will be compared between Hour 0 and Hour 3 at Visit 1 and Visit 2 to control for the effect of the substance on the subjects' levels of anxiety.
  The VAS ranges from 0 (no anxiety) to 100 mm (worst possible anxiety).
Change from Visit 1 (Day 0) in the score of visual analogue scale (VAS) on sadness at Visit 2 | From Visit 1 (Day 0) to Visit 2 (Day 7)
  The scores of the VAS-sadness will be compared between Hour 0 and Hour 3 at Visit 1 and Visit 2 to control for the effect of the substance on the subjects' levels of sadness.
  The VAS ranges from 0 (no sadness) to 100 mm (worst possible sadness).
Change from Visit 1 (Day 0) in the score of visual analogue scale (VAS) on fatigue at Visit 2 | From Visit 1 (Day 0) to Visit 2 (Day 7)
  The scores of the VAS-fatigue will be compared between Hour 0 and Hour 3 at Visit 1 and Visit 2 to control for the effect of the substance on the subjects' levels of fatigue.
  The VAS ranges from 0 (no fatigue) to 100 mm (maximum imaginable fatigue).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Neuromodulation, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
URL: https://www.osf.io